CLINICAL TRIAL: NCT03604081
Title: Effectiveness of Modified Constraint Induced Movement Therapy to Improve Lower Extremity Function in the Acute and Subacute Stroke Patients by Providing 1 Hour of Intense Massed Practice in the Form of Shaping or Task Practice, 7 Times Per Week for 2 Weeks.
Brief Title: Effectiveness of Modified Constraint Induced Movement Therapy to Improve Lower Extremity Function in the Acute and Subacute Stroke Patients by Providing 1 Hour of Intense Massed Practice in the Form of Shaping or Task Practice
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has encountered recruitment challenges.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-00773
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Stroke
Keywords: Constraint Induced Movement Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): One hour of intense massed practice of lower extremity either in the form of shaping or task practice
  Interventions: Other: CIMT
- Control Group (Placebo Comparator): Conventional physical therapy for 1 hour as per current standard of care that follows stroke clinical practice guideline.
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: CIMT — Intervention group will receive one hour of intense massed practice of lower extremity either in the form of shaping or task practice.
  Arms: Intervention Group
Other: Conventional Physical Therapy — 1 hour as per current standard of care that follows stroke clinical practice guideline.
  Arms: Control Group

SUMMARY:
This is a prospective randomized control trial of patients with unilateral impairment of the lower extremity after stroke. Patients will be randomized to intervention group and control group. Intervention group will receive one hour of intense massed practice of lower extremity either in the form of shaping or task practice. Control group will receive conventional physical therapy for 1 hour as per current standard of care that follows stroke clinical practice guideline.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 or older
* new ischemic stroke as revealed by CT scan or MRI of a brain or as per updated definition by American heart and American stroke association (Sacco et al., 2013)
* Manual muscle testing with grad of > 1+ in hip and knee joint musculature
* able to walk atleast 10 feet indoors with or without assistance and assistive device.
* Motivated to participate and some initiation of flexion and extension movement in hip, knee and ankle joints.
* Ability to follow visual/verbal instructions as assessed by a minimum score of 24/30 points on the minimental state examination
* Fairly intact sensation

Exclusion Criteria:

* Serious cardiac or pulmonary condition or other medical condition that make it difficult or risky to participate in intensive training
* Severe joint pain or degenerative disease to the musculoskeletal system of the lower extremity
* other neurological disease 4) problems with following instructions.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
Cycle time as measured by GAITRite. | 2 Weeks
  GAITrite is considered a gold standard for gait analysis. It consists of a mat with the sensors which are pressure sensitive and when patient ambulates on the mat the system measures parameters like step length, stride length, cycle time and velocity.
step length as measured by GAITRite. | 2 Weeks
  GAITrite is considered a gold standard for gait analysis. It consists of a mat with the sensors which are pressure sensitive and when patient ambulates on the mat the system measures parameters like step length, stride length, cycle time and velocity.
Stride length as measured by GAITRite. | 2 Weeks
  GAITrite is considered a gold standard for gait analysis. It consists of a mat with the sensors which are pressure sensitive and when patient ambulates on the mat the system measures parameters like step length, stride length, cycle time and velocity.
velocity as measured by GAITRite | 2 Weeks
  GAITrite is considered a gold standard for gait analysis. It consists of a mat with the sensors which are pressure sensitive and when patient ambulates on the mat the system measures parameters like step length, stride length, cycle time and velocity.

CONTACTS AND LOCATIONS:
Overall Officials: Nada Abou-Fayssal, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States